CLINICAL TRIAL: NCT07190781
Title: Development Platform Construction and Application Promotion of Drug-Eluting Stents for Intracranial Aneurysm Interventional Therapy
Status: Enrolling by invitation | Type: Observational
Sponsor: Xinjian Yang (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Beijing Chao Yang Hospital (Other); Peking University International Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Sponsor-Investigator, Xinjian Yang, Vice Director of the Neurosurgery Department, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Other Study IDs: KY-2025-231-03
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Aneurysm Unruptured

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Flow-Diverting Dense-Mesh Stent — Surface-Modified Flow-Diverting Dense-Mesh Stent for Mid-Term Follow-Up Study of Endovascular Embolization Therapy for Cerebral Aneurysms

SUMMARY:
This study is a post-marketing clinical study of the Lattice Flow-Diverting Dense-Mesh Stent. It plans to enroll 280 patients, who will be treated for unruptured intracranial aneurysms using the Lattice Flow-Diverting Dense-Mesh Stent. Patients will be followed up at 12 months after device implantation, and data including the Raymond classification of the target aneurysms, the occurrence of complications, and whether complications result in neurological deficit symptoms will be collected and assessed. Through the above indicators, the clinical safety and efficacy of the product will be evaluated.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria Aged 18 years or older; Patients diagnosed with unruptured intracranial aneurysms via CTA (Computed Tomographic Angiography), MRA (Magnetic Resonance Angiography), or DSA (Digital Subtraction Angiography); Patients treated with the Lattice Flow-Diverting Dense-Mesh Stent; Patients with 12-month follow-up records after treatment with the Lattice Flow-Diverting Dense-Mesh Stent; Patients whose aneurysms and parent arteries meet the indications for the Lattice Flow-Diverting Dense-Mesh Stent.

-

Exclusion Criteria:Patients with severe respiratory, circulatory, hepatic, renal diseases, or coagulation disorders; Patients whose target aneurysms are pseudoaneurysms, or aneurysms associated with arteriovenous malformations (AVMs) or Moyamoya disease; Patients with intracranial space-occupying lesions (such as intracranial tumors, abscesses, etc.), or those undergoing radiotherapy to the head; Patients currently participating in clinical trials of other drugs or medical devices; Patients with incomplete follow-up information 12 months after treatment with the Lattice Flow-Diverting Dense-Mesh Stent; Patients who express explicit disagreement (verbally or in writing) with participating in this study; Patients with parent artery stenosis greater than 50% that requires balloon angioplasty.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with unruptured intracranial aneurysms via CTA , MRA , or DSA
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Raymond-Roy Classification Scale | From Admission to the Hospital to 12 Months After the Completion of Surgical Treatment
  Raymond-Roy Classification Scale:
  Grade I: Complete occlusion; Grade II: Near-complete occlusion (with residual aneurysm neck or dog-ear sign); Grade III: Partial occlusion (with residual aneurysm sac).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No